CLINICAL TRIAL: NCT00886028
Title: "Phase II Study: Palliative Treatment With Liposomal Doxorubicin Plus Cisplatin for Patients With Malignant Pleural Mesothelioma "
Brief Title: Palliative Treatment With Liposomal Doxorubicin Plus Cisplatin for Patients With Malignant Pleural Mesothelioma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute of Cancerología (Other Government)
Responsible Party: Oscar Arrieta Rodríguez, CONACYT
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CB/304/06; 007/024/OMI
Record Dates: First submitted 2009-04-20; First posted 2009-04-22 (Estimated); Last update posted 2009-04-22 (Estimated); Status verified 2009-04

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: Malignant pleural mesothelioma; Liposomal doxorubicin; Progression free survival; Patients who received LD 60mg/m2 plus cisplatin 80 mg/m2 every 4 weeks for 6 cycles; Patients with epithelial, sarcomatoid or biphasic histological confirmed diagnosis of MPM
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — liposomal doxorubicin; Cisplatin

ARMS (1):
- Liposomal doxorubicin (Experimental): Thirty patients with MPM who received liposomal doxorubicin 60mg/m2 plus cisplatin 80 mg/m2 every 4 weeks for 6 cycles.
  Interventions: Drug: Liposomal doxorubicin; Drug: Cisplatin

INTERVENTIONS:
Drug: Liposomal doxorubicin — Liposomal doxorubicin 60 mg/m2 every 4 weeks for 6 cycles.
  Thirty patients with epithelial, sarcomatoid or biphasic histological confirmed diagnosis of MPM from the Instituto Nacional de Cancerología and the Instituto Nacional de Enfermedades Respiratorias were included to receive LD 60mg/m2 plus cisplatin 80 mg/m2 every 4 weeks for 6 cycles.
Drug: Cisplatin — Cisplatin 80 mg/m2 every 4 weeks for 6 cycles.
  Thirty patients with epithelial, sarcomatoid or biphasic histological confirmed diagnosis of MPM from the Instituto Nacional de Cancerología and the Instituto Nacional de Enfermedades Respiratorias were included to receive LD 60mg/m2 plus cisplatin 80 mg/m2 every 4 weeks for 6 cycles.

SUMMARY:
Liposomal doxorubicin consists on doxorubicin encapsulated in liposomes that are composed of phosphatidylcholine and cholesterol. Liposomal doxorubicin can extravasate into tumors with abnormal vascular endothelium but may not penetrate normal tissues lowering its toxicity and increasing its efficiency. Combining Liposomal doxorubicin with cisplatin could be an effective new chemotherapy treatment for malignant pleural mesothelioma .

Hypothesis:

Liposomal doxorubicin combined with cisplatin could increase response rates to chemotherapy, progression free survival and overall survival in patients with malignant pleural mesothelioma.

DETAILED DESCRIPTION:
Background:

Malignant pleural mesothelioma (MPM) is an invasive primary neoplasm associated with a rapid progression. It is usually diagnosed in the fifth to seventh decades of life, with a strong male predominance. 80% of the patients with MPM have a history of asbestos exposure. MPM develops only in 10% of the people with asbestos exposure, suggesting that other factors may be important in the development of this malignancy. MPM is classified into three pathological types: epithelial, sarcomatoid, and mixed. The epithelial type represents 50% of all the cases whether the sarcomatoid type the15%. Clinically the sarcomatoid type is related to a poorer prognosis compared with epithelial or mixed types MPM presents unique challenges with regard to diagnosis, staging, and treatment. Survival rates are approximately 6 months in patients without surgical treatment. 90% of the patients with MPM are not candidates for a surgical treatment because they arrived at advanced stages or with a poor lung function. In addition, surgery as a single modality has failed to improve survival, and several researches have explored the use of combined modality therapy incorporating radiation and chemotherapy. Given that the prognosis for patients with advanced MPM is poor regardless of the type of anticancer treatment, palliation of symptoms has been the primary goal. Chemotherapy remains the main palliative therapeutic modality, although either surgical intervention or local radiation therapy may be useful for the local control of pain or symptoms often associated with pleural fluid accumulation.

Most single chemotherapeutic agents have been tested in MPM obtaining response rates of < 20%. The impact of chemotherapy on the survival of patients with MPM remains uncertain. Platinum analogues have been extensively studied in MPM both single and combined regimens. There have been studies of patients with MPM treated with cisplatin 60 mg/m2 and doxorubicin 60 mg/m2 on day 1 with a 3 or 4 week interval demonstrating response rates of 20 to 25% with and overall survival of 10 months.

Liposomal doxorubicin (LD) consists on doxorubicin encapsulated in liposomes that are composed of phosphatidylcholine and cholesterol. LD can extravasate into tumors with abnormal vascular endothelium but may not penetrate normal tissues lowering its toxicity and increasing its efficiency. Combining LD with cisplatin could be an effective new chemotherapy treatment for MPM.

Objective:

Increase chemotherapy response rates, progression free survival and overall survival in patients with MPM treated with LD plus cisplatin as a palliative treatment for MPM.

Methods:

We conducted a prospective analytical study between September 2006 and April 2009. Thirty patients with epithelial, sarcomatoid or biphasic histological confirmed diagnosis of MPM from the Instituto Nacional de Cancerología and the Instituto Nacional de Enfermedades Respiratorias were included to receive LD 60mg/m2 plus cisplatin 80 mg/m2 every 4 weeks for 6 cycles. During the first cycle of chemotherapy, a scintigraphic image study was done with LD labeled with Tc-99m (LD-Tc-99m). The imaging study (SPECT/CT) was done 1h after administration to evaluate biodistribution and accumulation of LD-Tc-99m in tumoral tissue. Patients were evaluated by a surgeon after 2 cycles of chemotherapy, if surgery was not possible, chemotherapy continued until tumor progression. Clinical and biochemical evaluations were obtained before chemotherapy administration. An axial computed tomography was requested before chemotherapy and every 2 months in the first 6 months and every 4 months during following 2 years. Treatment response was according to RECIST criteria and toxicity was evaluated with National Cancer Institute Common Toxicity Criteria version 3.0. The statistical analysis was made using SPSS v.10 software. For descriptive purposes, continuous variables were summarized as arithmetic means, medians, and standard deviations; and categorical variables with 95% confidence intervals. Disease-free progression and over-all survival were evaluated by Kapplan-Meier.

ELIGIBILITY:
Inclusion Criteria:

* Patients with epithelial, sarcomatoid or biphasic histological confirmed diagnosis of MPM from the Instituto Nacional de Cancerología and the Instituto Nacional de Enfermedades Respiratorias
* ECOG functional status 0 or 2
* No renal function alteration (GFR >50%)
* No hepatic function alteration
* Leucocytes more than 2,000/mcl
* Hemoglobin more than 10mg/dL
* Platelets more than 100,000/mcl

Exclusion Criteria:

* Patients who had received previous chemotherapy for MPM
* Patients who do not accept the treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2006-09; Primary Completion 2009-04 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 12 months
Over-all survival | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Estrada Lobato, M.D., Study Chair — National Institute of Cancerología; Luis Alberto Medina Velázquez, PhD., Study Chair — Laboratorio de Enseñanza Virtual y Ciberpsicología. Facultad de Psicología. UNAM; Elena Arechaga Ocampo, PhD., Study Chair — National Institute of Cancerología; Victoria López Rodrígez, Q.F.B., Study Chair — National Institute of Cancerología; Luisa Geraldine Villanueva Rodríguez, M.D, Study Chair — National Institute of Canerología; Miguel Angel Ríos Trejo, M.D., Study Chair — National Institute of Cancerología
Locations (1):
- National Institute of Cancerología, Mexico City, Mexico City, Mexico

REFERENCES:
- [Derived] Arrieta O, Medina LA, Estrada-Lobato E, Hernandez-Pedro N, Villanueva-Rodriguez G, Martinez-Barrera L, Macedo EO, Lopez-Rodriguez V, Motola-Kuba D, Corona-Cruz JF. First-line chemotherapy with liposomal doxorubicin plus cisplatin for patients with advanced malignant pleural mesothelioma: phase II trial. Br J Cancer. 2012 Mar 13;106(6):1027-32. doi: 10.1038/bjc.2012.44. Epub 2012 Feb 21. PMID 22353806